CLINICAL TRIAL: NCT00115583
Title: The Contribution of Endothelin to Vasoreactivity in Atherosclerotic Coronary Arteries
Brief Title: The Contribution of Endothelin to Vasomotor Function in Diseased Coronary Arteries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Peter A. Ganz, Brigham & Women's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 1999-P-003104; P01HL048743 (NIH)
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Atherosclerosis, Coronary
MeSH Terms: conditions — Coronary Artery Disease | interventions — cyclo(Trp-Asp-Pro-Val-Leu)

INTERVENTIONS:
Drug: Drug Infusion (BQ-123)

SUMMARY:
The purpose of the study is to assess the importance of a substance called endothelin. Endothelin is produced by coronary arteries. This study examines this substance to determine whether it has an effect on controlling blood flow in coronary arteries. When these arteries release too much endothelin, the blood flow to the heart muscle is reduced and this may be important in heart conditions. This protocol examines an investigational drug called BQ-123 to see if it blocks the effect of endothelin. We assess the blood flow in the coronaries and evaluate the effects of BQ-123. It is anticipated that this endothelin blocker will open up coronary arteries and increase the blood flow to the heart.

DETAILED DESCRIPTION:
There are many substances that influence the diameter of the coronary artery and a number of these are actually released by the lining of the coronary arteries (referred to as the endothelium). Over the past 15 years, our laboratory has been instrumental in establishing the role of endothelium-released relaxing factors which relax (open) the coronary arteries. We are now focussing our attention on factors which constrict the coronary artery, in particular a substance called endothelin-1 (ET-1). This potent constrictor substance has been found to accumulate at coronary artery sites which may produce unstable angina (ie the culprit lesion or stenosis). Hence ET-1 may produce localized constriction of a coronary stenosis thereby further narrowing the remaining lumen and cutting off blood flow to the heart muscle and thus leading to unstable angina.

If ET-1 is important in the development of unstable angina, then medications which inhibit the effects of ET-1 should improve the condition. To achieve a blockade of ET-1, inhibitors of the two receptors (ET-A and ET-B) responsible for ET-1's action must be administered. Animal and human studies have demonstrated that a blockade of the ET-A receptor by the new antagonist, BQ-123, inhibits most of the ET-1 induced constrictor response. BQ-123 has been safely administered systemically by intravenous infusion and locally in the human forearm where it produces dilation of the forearm arteries. It has not been previously administered into human coronary arteries.

Consented patients whose routine diagnostic angiogram shows suitable anatomy (i.e., normal angiogram for the control group, or one/two vessel coronary artery disease with an identifiable culprit stenosis) will have placement of a coronary artery angiographic catheter. Placement of this catheter does not require an additional puncture of an artery (already performed in the routine diagnostic angiogram).

The angiographic catheter allows visualization of the internal diameter of the coronary arteries by the injection of a radiographic contrast with the image being recorded on a cine film. Specialized imaging machines will measure the diameter of the vessel.

Through the angiographic catheter, an infusion catheter (by which the drugs can be administered) and a coronary Doppler flow wire are placed in the coronary artery. The latter instrument is a well-established tool for measuring coronary blood flow.

After establishing baseline values for heart rate, blood pressure, culprit stenosis internal diameter and coronary blood flow, the following sequential intracoronary infusions will be undertaken:

1. Infusion of the endothelin antagonist, BQ-123, over a 60 minute period. This inhibitor requires up to 60 minutes exerting a full effect;
2. Adenosine bolus injection, to assess the vasodilation capacity of the small coronary arteries; and
3. Nitroglycerin bolus injection, to assess the maximal vasodilation capacity of the large coronary arteries.

At 5, 15, 30, 45, and 60 minutes of endothelin antagonist infusion, and immediately after the bolus injections, the above parameters will be reassessed. It is anticipated that this research protocol will be completed within 90 minutes.

Following the research protocol, the patient will undergo appropriate coronary intervention as dictated by the clinical situation. If coronary atherectomy is required for clinical indications, then the specimen extracted by this procedure will be sent for specific analysis of endothelin-1 content. A correlation between the amount of endothelin at the culprit stenosis and the response to the endothelin antagonist can then be examined. In cardiac transplant recipients, endomyocardial biopsies are also routinely obtained for clinical purposes at the time of catheterization. One of these specimens will be used for ET-1 immunoreactivity analysis. A total of 2 teaspoons of blood will be taken and frozen for analysis.

ELIGIBILITY:
Inclusion Criteria:

Adult men and women between the ages of 18 to 75 years will be enrolled and categorized into one of 4 groups. The categories are defined below:

* Control patients characterized by chest pain and angiographically normal coronary arteries.
* Chronic stable angina patients who describe a history of exertional chest pain which is unchanged in frequency over the preceding month, and who have at least a 70% stenosis in a coronary artery.
* Unstable angina patients who describe chest pain at rest or with minimal exertion over the preceding 2 weeks, and who have an identifiable culprit stenosis in a coronary artery.
* Cardiac transplant recipients who are undergoing routine annual surveillance cardiac catheterization.

Exclusion Criteria:

Patients with the following will be excluded from the study:

* Angiographic exclusion criteria: *Left main coronary artery disease or severe triple vessel disease; *Unstable angina without any identifiable culprit lesion.
* Severe left ventricular dysfunction (ejection fraction < 40%) or clinical cardiac failure.
* Nitroglycerin required in the preceding 4 hours prior to the investigation.
* Severe renal, hepatic or hematologic abnormalities.
* Inability to obtain written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1998-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in minimum luminal diameter from baseline assessed by Quantitative Angiography
Coronary Flow Reserve (max/basal CBFV) assessed by coronary Doppler Wire
Correlation between the change in culprit epicardial artery stenosis MLD and atherectomy specimen ET-1 content assessed by immunochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Ganz, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States